CLINICAL TRIAL: NCT06460389
Title: Comparison of Visual Outcomes After Extended Depth of Focus Intraocular Lens Implantation with and Without Digital Assistance
Brief Title: Visual Outcomes After Extended Depth of Focus Intraocular Lens Implantation with and Without Digital Assistance
Status: Recruiting | Type: Observational
Sponsor: Democritus University of Thrace (Other)
Responsible Party: Principal Investigator, Georgios Labiris, Professor (Associate) of Democritus University of Thrace, Democritus University of Thrace
Other Study IDs: ES6/Th11/14-03-2024
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Presbyopia; Pseudophakia; Cataract; Refractive Errors
Keywords: pseudophakic presbyopic correction; extended depth of field intraocular lenses; visual curve; visual acuity
MeSH Terms: conditions — Presbyopia; Pseudophakia; Cataract; Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Insertion of an extended depth of focus intraocular lens with digital assistance: Participants that underwent uncomplicated IOL implantation of an extended depth of focus intraocular lens with digital assistance
  Interventions: Diagnostic Test: Visual Acuity Assessment
- Insertion of an extended depth of focus intraocular lens without digital assistance: Participants that underwent uncomplicated IOL implantation of an extended depth of focus intraocular lens without digital assistance
  Interventions: Diagnostic Test: Visual Acuity Assessment

INTERVENTIONS:
Diagnostic Test: Visual Acuity Assessment — Uncorrected visual acuity for nine distances (25, 28, 33, 40, 50, 60, 100, 200, 300 cm) examination via a Democritus Digital Acuity & Reading Test (DDART).

SUMMARY:
The primary objective of this study is to compare the postoperative visual acuity curves of patients that underwent one of the following surgical procedures: Insertion of an extended depth of focus intraocular lens with digital assistance and insertion of an extended depth of focus intraocular lens without digital assistance.

DETAILED DESCRIPTION:
This is a prospective, comparative study of 60 patients diagnosed with grade 2 cataracts (according to LOCS III) that underwent one of the following surgical procedures: Insertion of an extended depth of focus intraocular lens with digital assistance and insertion of an extended depth of focus intraocular lens without digital assistance.

In these patients, a comparison of postoperative visual acuity curves of both groups will be conducted. Visual acuity curves will be designed using the validated digital optotype Democritus Digital Acuity & Reading Test (DDART). Assessment of visual acuity will be performed at 9 different distances (25, 28, 33, 40, 50, 60, 100, 200, 300 cm). Overall visual acuity curves and the area under the curve will be formed through the application as the primary means of evaluating visual capacity. Additionally, the degree of subjective satisfaction of the patient will be evaluated through an interview (NEI-VFQ 25). All examinations will be conducted according to standard clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of grade 2 cataracts (according to LOCS III)
* age >45 years.

Exclusion Criteria:

* Inability to understand the Greek language and respond to the interview
* conditions of the posterior or corneal segment
* glaucoma
* previous intraocular surgery

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants that underwent Extended Depth of Focus Intraocular Lens Implantation With and Without Digital Assistance.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Visual acuity assessment | 4 months
  Visual acuity assessment in 9 focal points using DDART chart
Area of the curve (AOC) assessment | 4 months
  Calculation of the AOC as a visual outscome measure
the degree of subjective satisfaction of the patient | 4 months
  the degree of subjective satisfaction of the patient will be evaluated through an interview (NEI-VFQ 25)

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Labiris, Study Chair — Democritus University of Thrace
Locations (1):
- Department of Ophthalmology, University Hospital of Alexandroupolis, Alexandroupoli, Evros, Greece

IPD SHARING:
Plan to Share IPD: No